CLINICAL TRIAL: NCT01221207
Title: Instant Total Contact Cast to Heal Diabetic Foot Ulcers
Acronym: ITCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Larry Lavery, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTSW - 7R01DK074483-04
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic foot ulcers; casting; wound care
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Device - Total Contact Cast (TCC) (Active Comparator): A total contact cast (TCC) is a special cast technique that is used to take the pressure and shear stress off the ulcer to assist in the healing.
  Interventions: Device: Total Contact Cast
- Removable Cast Walker (RCW) (Active Comparator): The removable cast walker (RCW) is a commercial product that is similar to a cast. It is secured with Velcro straps around the foot and leg and it is also effective at removing the pressure and shear stress on the foot.
  Interventions: Device: Removable Cast Walker (RCW)
- Instant Total Contact Cast (ITCC) (Active Comparator): The instant total contact cast (ITCC) is a technique that uses the removable cast walker, but secures it so it cannot be removed between clinic visits and evaluation by the subject or the physician.
  Interventions: Device: Instant Total Contact Cast (ITCC)

INTERVENTIONS:
Device: Total Contact Cast — A total contact cast (TCC) is a special cast technique that is used to take the pressure and shear stress off the ulcer to assist in the healing.
  Arms: Device - Total Contact Cast (TCC)
Device: Instant Total Contact Cast (ITCC) — The instant total contact cast (ITCC) is a technique that uses the removable cast walker, but secures it so it cannot be removed between clinic visits and evaluation by the subject or the physician.
  Arms: Instant Total Contact Cast (ITCC)
Device: Removable Cast Walker (RCW) — The removable cast walker (RCW) is a commercial product that is similar to a cast. It is secured with Velcro straps around the foot and leg and it is also effective at removing the pressure and shear stress on the foot.
  Arms: Removable Cast Walker (RCW)

SUMMARY:
Aim 1. To compare the effectiveness of total contact casts (TCC), removable cast walkers (RCW) and instant total contact casts (ITCC) to heal diabetic foot ulcers in a 20 week randomized clinical trial of 225 patients in community care in three university medical center diabetes clinics.

Aim 2. To compare the frequency of complications such as soft tissue and bone infections, iatrogenic wounds, falls and fall related injuries, and amputations among patients treated with TCC, ITCC and RCW to heal diabetic foot ulcers.

Aim 3. To compare patient compliance and level of activity among TCC, ITCC, RCW treatment groups. Using computerized activity monitors which time-stamp each step, we will evaluate both degree and magnitude of activity between groups.

Aim 4. To evaluate the cost of diabetic foot ulcer-related treatment and complications during the course of therapy.

DETAILED DESCRIPTION:
This is an investigator blinded randomized, controlled clinical trial with three parallel treatment groups of 75 adult outpatients with diabetes mellitus and a foot ulcer. The study will be conducted at five university affiliated medical centers in Arizona and Texas. The study participants and nurse coordinator will not be blinded to the treatment after randomization. Investigators will be blinded to treatment group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years old or older
* One or more foot ulcers without clinical evidence of osteomyelitis
* Diagnosis of Diabetes Mellitus
* University of Texas Grade 1A-B, 2A-B or 3A-B
* ABI >0.5
* Spanish-speaking subjects will be eligible to participate

Exclusion Criteria:

* Active Charcot Arthropathy
* ABI <0.5
* Gangrene, active infection
* Unable to keep research appointments
* Wide spread malignancy or systemically immunocompromising disease
* Alcohol or substance abuse within 6 months
* Unreliable, unwilling or unable to comprehend informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - Parkland Health & Hospital Systems, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Scott & White, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Instant Total Contact Cast (ITCC) | Device - Total Contact Cast (TCC) | Removable Cast Walker (RCW)
Started | 75 | 75 | 75
Completed | 43 | 66 | 54
Not Completed | 32 | 9 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Instant Total Contact Cast (ITCC) | Device - Total Contact Cast (TCC) | Removable Cast Walker (RCW) | Total
Number analyzed (Participants) | 75 | 75 | 75 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.77 (11.99) | 52.61 (10.73) | 54.32 (12.61) | 53.59 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 15 | 46
  Male | 56 | 63 | 60 | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 43 | 33 | 34 | 110
  African American | 6 | 13 | 12 | 31
  Native American | 1 | 2 | 3 | 6
  Hispanic | 25 | 27 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve Full Wound Healing.
Description: We will evaluate wounds at each clinical visit. An ulcer will be considered "healed" when it is fully epithelialized with no drainage.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Instant Total Contact Cast (ITCC) | Device - Total Contact Cast (TCC) | Removable Cast Walker (RCW)
Number analyzed (Participants) | 75 | 75 | 75
Participants | 35 | 63 | 37

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Instant Total Contact Cast (ITCC) | Device - Total Contact Cast (TCC) | Removable Cast Walker (RCW)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 7/75 | 12/75 | 13/75
Other Adverse Events (participants affected / at risk) | 30/75 | 38/75 | 48/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Instant Total Contact Cast (ITCC) (N=75) | Device - Total Contact Cast (TCC) (N=75) | Removable Cast Walker (RCW) (N=75)
Foot related readmission (Infections and infestations) | 7 (9) | 12 (14) | 13 (16)
Non-foot related readmission (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Instant Total Contact Cast (ITCC) (N=75) | Device - Total Contact Cast (TCC) (N=75) | Removable Cast Walker (RCW) (N=75)
Soft tissue infection (Infections and infestations) | 6 (10) | 8 (12) | 12 (13)
Bone infection (Infections and infestations) | 6 (17) | 5 (10) | 7 (10)
New foot ulcer (Skin and subcutaneous tissue disorders) | 17 (30) | 23 (57) | 28 (57)
Mechanical fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (3)
Minor amputation of foot (Surgical and medical procedures) | 1 (2) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No